CLINICAL TRIAL: NCT04344223
Title: Effects of Stabilization Shoes on Balance and Walking. A Cross-over, Controlled, Randomized Single Blind Study.
Brief Title: Effect of Stabilization Shoes on Balance in Elderly
Acronym: BALAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Burgundy (Other)
Responsible Party: Principal Investigator, Nicolas Babault, Principal investigator, University of Burgundy
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CEP2001
Record Dates: First submitted 2020-04-01; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Elderly
Keywords: Postural Balance; Accidental Falls; Footwear; Stability; Force platform; Unipedal stance; Bipedal stance; Shoe

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data and statistical analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental balance shoes (Experimental): Tests and familiarization phases with experimental balance shoes (Axis Comfort Development®)
  Interventions: Device: Balance Shoe
- Personal shoes (Active Comparator): Same tasks than the condition "Experimental balance shoes" but realized with personal shoes (own personal shoes of subjects)
  Interventions: Device: Personal Shoe

INTERVENTIONS:
Device: Balance Shoe — Use of experimental balance shoes for carrying out the tests along the three sessions and one of the two familiarization phases
  Other Names: Axis Comfort Development® Experimental Balance shoes
  Arms: Experimental balance shoes
Device: Personal Shoe — Use of Personal shoes (the same for each session) for carrying out the tests along the three sessions and one of the two familiarization phases
  Other Names: Own personal shoes of subjects
  Arms: Personal shoes

SUMMARY:
Movement during everyday activities most often requires stable posture. Postural control corresponds to a complex motor ability to maintain / re-establish balance and orient one's body in the environment. Postural stability and equilibrium deteriorate with age. More than 30% of people over 65 years old fall per year. Falls represent 90% of hip fractures and sometimes result in lasting psychological effects. Shoes are our direct link between the ground and our feet. Wearing shoes plays a major role in postural control. The characteristics of shoes usually worn by elderly people are identified with those of shoes known to be 'dangerous'. In order to improve stability and reduce the risk of falling for the elderly, Axis-Comfort Development® has developed "experimental balance shoes". Their shoes have technical characteristics presented in the scientific literature as beneficial for postural stability.

Therefore, the aim of this study was to investigate the effects of wearing experimental balance shoes on postural balance compared with the people's own shoes. We assumed that postural balance would be improved by experimental balance shoes in an acute way and improved by a familiarization phase.

This was a controlled, randomized, blind and cross-over study. three sessions were held in our center, each time interspersed with a phase of familiarization at home (7 to 10 days) during which the people had to wear either the experimental balance shoes or their own personal shoes. 21 volunteers in total participated in this study, all between 65 and 75 years old. Five tests were presented randomly for each session and all tests were carried out on a Huber 360 ® (LPG System, France) stabilometric platform. The mains criteria were static equilibrium on one foot and two feet (with eyes open and closed) and secondary criteria were stride frequency during the walk on the spot and stability limits.

An improvement of these multiple criteria during the different sessions would be proof of the positive effect of experimental balance shoes on postural balance in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 65 to 75 years old
* Healthy subjects
* Having given their written informed consent

Exclusion Criteria:

* Subject who has fallen during the six months prior to the study.
* Subject who moves with walking aids.
* Subject with severe balance problems or unable to stand up without help
* Subject who takes sedatives or sleeping pills
* Subject with neurological disease (dizziness including turning dizziness, multiple sclerosis, Parkinson's, etc.)
* Subject with history of heart attack
* Subject who is short of breath when inactive.
* Subject who has pains limiting walking and standing
* Subject who takes neuroleptics except Anti-depressors if the treatment is long-standing and well-balanced.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Assessing change of the displacement surface of the center of pressure between the three sessions during static balance on a foot with open eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Surface of the displacement of the centre of pressure (Value in square millimeters, mm²) during 30 seconds was measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change of the length of the displacement of the centre of pressure between the three sessions during static balance on a foot with open eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Length of the displacement of the centre of pressure (Value in millimeters, mm) during 30 seconds was measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change of the number of rebalancing gestures between the three sessions during static balance on a foot with open eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Number of rebalancing gestures (with the foot or with the hand during test) during 30 seconds was measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change of the displacement surface of the center of pressure between the three sessions during static balance on two feet open eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Surface of the displacement of the centre of pressure (Value in square millimeters, mm²) during 50 seconds was measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change of the length of the displacement of the centre of pressure between the three sessions during static balance on two feet open eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Length of the displacement of the centre of pressure (Value in millimeters, mm) during 50 seconds was measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change of the average speed of the displacement of the centre of pressure between the three sessions during static balance on two feet open eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Average speed of the displacement of the centre of pressure (Value in millimeters per second, mm/s) during 50 seconds was measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change of the number of rebalancing gestures between the three sessions during static balance on two feet open eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Number of rebalancing gestures (with the foot or with the hand during test) during 50 seconds was measured on a Huber 360 ® (LPG System, France) force platform.

SECONDARY OUTCOMES:
Assessing change in walking capacity between the three sessions | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Walk at the pace following the change of the Left (on right foot and left leg detached) and Right (opposite) visuals on the platform screen for 50 seconds. Subjects were asked to lift their feet using enough hip flexion to bring the foot halfway up the support leg. The expected number of strides was around 96. Measured on a Huber 360 ® (LPG System, France) force platform (number of strides).
Assessing change in stability limits between the three sessions at 0° | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Maximal displacement of the centre of pressure at 0°. 8 seconds to go as far as possible (Value in degrees, °). Measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change in stability limits between the three sessions at 45° | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Maximal displacement of the centre of pressure at 45°. 8 seconds to go as far as possible (Value in degrees, °). Measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change in stability limits between the three sessions at 90° | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Maximal displacement of the centre of pressure at 90°. 8 seconds to go as far as possible (Value in degrees, °). Measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change in stability limits between the three sessions at 135° | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Maximal displacement of the centre of pressure at 135°. 8 seconds to go as far as possible (Value in degrees, °). Measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change in stability limits between the three sessions at 180° | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Maximal displacement of the centre of pressure at 180°. 8 seconds to go as far as possible (Value in degrees, °). Measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change in stability limits between the three sessions at 225° | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Maximal displacement of the centre of pressure at 225°. 8 seconds to go as far as possible (Value in degrees, °). Measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change in stability limits between the three sessions at 270° | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Maximal displacement of the centre of pressure at 270°. 8 seconds to go as far as possible (Value in degrees, °). Measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change in stability limits between the three sessions at 315° | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Maximal displacement of the centre of pressure at 315°. 8 seconds to go as far as possible (Value in degrees, °). Measured on a Huber 360 ® (LPG System, France) force platform.
Subjective assessment of the comfort linked to the wearing of the experimental balance shoes | Measured after wearing experimental balance shoes for a week (familiarization's period)
  The question was : "How do you feel in general wearing Balance Shoes?" with 4 predefined answers : (1) "Very comfortable" ; (2) "Comfortable" ; (3)"Normal" and (4) "Uncomfortable". Questionary was anonymous
Subjective assessment of the aesthetics linked to wearing of the experimental balance shoes | Measured after wearing experimental balance shoes for a week (familiarization's period)
  The question was : "How do you find the aesthetics of Balance Shoes?" with 4 predefined answers : (1) "To my liking" ; (2) "Correct" ; (3)"Not to my liking" and (4) "No opinion". Questionary was anonymous
Subjective assessment of the stability linked to wearing of the experimental balance shoes | Measured after wearing experimental balance shoes for a week (familiarization's period)
  The question was : "Did you feel more stable wearing Balance Shoes?" with 2 predefined answers : (1) "Yes" ; (2) "No". Questionary was anonymous
Subjective assessment of the safety linked to wearing of the experimental balance shoes | Measured after wearing experimental balance shoes for a week (familiarization's period)
  The question was : "Did you feel safer wearing Balance Shoes?" with 2 predefined answers : (1)"Yes" ; (2) "No". Questionary was anonymous
Assessing change of the displacement surface of the center of pressure between the three sessions during static balance on two feet closed eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Surface of the displacement of the centre of pressure (Value in square millimeters, mm²) during 50 seconds was measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change of the length of the displacement of the centre of pressure between the three sessions during static balance on two feet closed eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Length of the displacement of the centre of pressure (Value in millimeters, mm) during 50 seconds was measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change of the average speed of the displacement of the centre of pressure between the three sessions during static balance on two feet open eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Average speed of the displacement of the centre of pressure (Value in millimeters per second, mm/s) during 50 seconds was measured on a Huber 360 ® (LPG System, France) force platform.
Assessing change of the number of rebalancing gestures between the three sessions during static balance on two feet open eyes | Measure during the three sessions and for both conditions (balance or personal). 1 minute recovery between tests. 7 to 10 days between the three sessions (familiarization). Test appearance order is random for each session
  Number of rebalancing gestures (with the foot or with the hand during test) during 50 seconds was measured on a Huber 360 ® (LPG System, France) force platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Expertise de la Performance - Université de Bourgogne, Dijon, Côte d'Or, France

IPD SHARING:
Plan to Share IPD: No